CLINICAL TRIAL: NCT01939782
Title: Metabolic Clock Gene Expression in Peripheral Blood Cells During Fasting and After Food Intake in the Breakfast in Type 2 Diabetic Patients
Brief Title: Metabolic Clock Genes During Fasting and After Food Intake in Type 2 Diabetics
Acronym: MCG-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof. Daniela Jakubowicz MD, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0102-13-WOMC
Record Dates: First submitted 2013-09-02; First posted 2013-09-11 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
Keywords: Metabolic CLock Genes (MCG); Type 2 Diabetes (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type 2 diabetic patients (T2D) (Experimental): In type 2 diabetic patients (T2D), the investigators will evaluate the metabolic clock gene expression in PBC and serum glucose, insulin, triglycerides, free fatty acids (FFA), cortisol intact GLP-1, triglycerides ,cortisol, plasma free fatty acids (FFA l and DPP4 plasma activity in two different occasions:
  1. No Breakfast (NoB): fasting until lunch at 12:00
  2. Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00 In both occasions the blood samples for glucose and insulin, cortisol and intact GLP-1 will be taken after overnight fast at 8:30 and thenat 8:30, 9:00, 10:30, 12:00, 12:30, 14:00 and 15:30. The samples for clock genes and for DPP4 plasma activity will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2 h after lunch).
  Interventions: Other: No Breakfast (NoB); Other: Yes Breakfast (YesB)
- Healthy No Diabetics (Active Comparator): In healthy No Diabetics,: the investigators will evaluate the metabolic clock gene expression in PBC and serum glucose, insulin, triglycerides, free fatty acids (FFA), cortisol intact GLP-1, triglycerides ,cortisol, plasma free fatty acids (FFA l and DPP4 plasma activity in two different occasions:
  1. No Breakfast (NoB): fasting until lunch at 12:00
  2. Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00 In both occasions the blood samples for glucose and insulin, cortisol and intact GLP-1 will be taken after overnight fast at 8:30 and thenat 8:30, 9:00, 10:30, 12:00, 12:30, 14:00 and 15:30. The samples for clock genes and for DPP4 plasma activity will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2 h after lunch).
  Interventions: Other: No Breakfast (NoB); Other: Yes Breakfast (YesB)

INTERVENTIONS:
Other: No Breakfast (NoB) — In both occasions the blood samples for glucose and insulin, cortisol triglycerides and intact GLP-1 will be taken after overnight fast at 8:30 and thenat 8:30, 9:00, 10:30, 12:00, 12:30, 14:00 and 15:30. The samples for clock genes and for DPP4 plasma activity will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2 h after lunch).
  Other Names: NoB
Other: Yes Breakfast (YesB) — In both occasions the blood samples for glucose and insulin, cortisol, triglycerides and intact GLP-1 will be taken after overnight fast at 8:30 and then at 8:30, 9:00, 10:30, 12:00, 12:30, 14:00 and 15:30. The samples for clock genes and for DPP4 plasma activity will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2 h after lunch).
  Other Names: YesB

SUMMARY:
This study is undertaken to explore whether compared to extension of overnight fast until lunch versus the breakfast consumption influence the oscillation of the metabolic clock gene expression in peripheral blood cells (PBC), at noon and after isocaloric lunch in type 2 diabetic patients.

DETAILED DESCRIPTION:
Most of our metabolic function is controlled by metabolic clock genes that regulate glucose, lipid metabolism and several other circadian metabolic pathways involved in insulin resistance obesity and type 2 diabetes. The main group of clock genes resides in the SCN nuclei and is synchronized by light/dark signals. However similar clock oscillators called peripheral clocks are found in almost all tissues, including in the liver, heart, kidney, intestine, skeletal muscles, and adipocytes and in peripheral blood cells (PBC). The peripheral clocks, and specially those metabolic clock genes, seem to be controlled mainly by food cues.

The time of food intake synchronize simultaneously and in parallel way almost all the peripheral metabolic clock genes including those expressed and in peripheral blood cells (PBC) i.e. leucocytes, monocytes; allowing to explore the oscillation of the metabolic clock gene expression of the whole body by assessing its expression in the PBC. Impaired oscillation of the metabolic clock gene mRNA expression was found in diabetic animal models and in patients with type 2 diabetes and were inversely correlated with HbA1c.

In support of these finding we reported that high calorie breakfast with reduced dinner improved insulin sensitivity and weight loss rate among obese subjects, while in type 2 diabetic patients the high calorie breakfast was associated with improvement of HbA1c.

Moreover, recently was shown that very short time (only 120 min) after food intake in the breakfast, was sufficient to reset the expression of the circadian clock genes.

This study is undertaken to explore whether compared to extension of overnight fast until lunch versus the breakfast consumption influence the oscillation of the metabolic clock gene expression in peripheral blood cells (PBC), at noon and after isocaloric lunch in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR PATIENTS WITH TYPE 2 DIABETES

1. Type 2 diabetic patients
2. HbA1C > 6.5%
3. Duration of diabetes: 0.5 to 30 years
4. Subjects ≥ 26 and ≤ 65 years of age
5. BMI: > 26 kg/m2
6. All oral antidiabetic treatments and will be allowed, not insulin treatment
7. Normal liver and kidney function
8. Normal thyroid function
9. Stable physical activity pattern during the three months immediately preceding study
10. No metabolic disease other than diabetes
11. Usually wakes up between 06:00 and 07:00 and goes to sleep between 22:00 and 24:00.
12. Normal TSH and FT4 levels
13. No shift work within 5 years of the study
14. Did not cross time zones within 1 month of the study
15. Acceptable health beside diabetes based on interview, medical history, physical examination, and laboratory tests
16. Read and understood the informed consent form and signed it voluntarily

INCLUSION CRITERIA FOR HEALTHY NON-DIABETIC PATIENTS

1. Healthy non diabetic, and not known as diabetic
2. Fating glucose <100 mg/dl
3. HbA1C <5.7 %
4. Not taking any antidiabetic drugs
5. Subjects ≥ 26 and ≤ 65 years of age
6. BMI: <26 kg/m2
7. Normal liver and kidney function
8. Normal TSH and FT4 levels
9. Usually wakes up between 06:00 and 07:00 and goes to sleep between 22:00 and 24:00.
10. No shift work within 5 years of the study
11. Did not cross time zones within 1 month of the study
12. Acceptable health based on interview, medical history, physical examination, and laboratory tests
13. Read and understood the informed consent form and signed it voluntarily

Exclusion Criteria:

EXCLUSION CRITERIA FOR ALL 2 GROUPS (HEALTHY AND DIABETICS)

1. Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, malignant disease
2. Type 1 diabetes
3. Treatment with Insulin
4. Serum creatinin level > 1.5 mg/dl
5. Pregnancy or lactation
6. Illicit drug abuse or alcoholism
7. Subjects taking anoretic drugs during the month immediately prior to study
8. Subjects on steroid treatment
9. Subjects known by the principal investigator to be unable to cooperate for any reason.
10. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)
11. Night or rotating shift work
12. Jet lag during the 2 week period immediately prior to study onset

Ages: 26 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Metabolic Clock Gene Expression in Peripheral Blood Cells(PBC), | Blood samples for the clock genes will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2h after lunch)
  In all subjects the the blood samples for metabolic clock gene expression in PBC will be evaluated in PBC in two different occasions Fasting No Breakfast (NoB): fasting until lunch at 12:00 Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00 In both occasions the blood samples for the clock genes will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2 h after lunch)

SECONDARY OUTCOMES:
Serum glucose insulin and intact GLP-1 levels | Blood samples for glucose insulin and intact GLP-1 levels will be taken after overnight fast at 8:30 and then at 9:00, 10:30 , 12:00, 12:30, 14:00 and 15:30
  In all subjects the the blood samples for serum glucose insulin and intact GLP-1 levels will be evaluated, in two different occasions:
  No Breakfast (NoB): fasting until lunch at 12:00 Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00 In both occasions the blood samples for glucose and insulin will be taken after overnight fast at 8:00 and then every hour until 15:30.
Serum Triglycerides and Free Fatty Acids | Blood samples for Triglycerides and Free Fatty Acids will be taken after overnight fast at 8:30 and then at 9:00, 10:30 , 12:00, 12:30, 14:00 and 15:30
  In all subjects the the blood samples for serum Triglycerides and Free Fatty Acids plasma levels will be evaluated, in two different occasions No Breakfast (NoB): fasting until lunch at 12:00 Yes Breakfast (YesB): eating breakfast at Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00
DPP4 plasma activity | Blood samples for DPP4 plasma activity will be taken after overnight fast at 8:30, before lunch at 12:00 and at 15:30
  In all subjects the the blood samples for DPP4 plasma activity will be evaluated in PBC in two different occasions No Breakfast (NoB): fasting until lunch at 12:00 Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00 In both occasions the blood samples for DPP4 plasma activity will be taken at 8:30, 12:00 (before lunch) and at 15:30 (3 1/2 h after lunch)
Serum Cortisol | Blood samples for Cortisol will be taken after overnight fast at 8:30 and then at 9:00, 10:30, 12:00, 12:30, 14:00 and 15:30
  In all subjects the the blood samples for serum Cortisol will be evaluated, in two different occasions No Breakfast (NoB): fasting until lunch at 12:00 Yes Breakfast (YesB): eating breakfast at Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00 Yes Breakfast (YesB): eating breakfast at Yes Breakfast (YesB): eating breakfast at 8:30 and lunch at 12:00

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Diabetes Unit E. Wolfson Medical Center. Tel Aviv University
Locations (1):
- Daniela Jakubowicz MD, Holon, N/A = Not Applicable, Israel

REFERENCES:
- [Derived] Jakubowicz D, Wainstein J, Landau Z, Raz I, Ahren B, Chapnik N, Ganz T, Menaged M, Barnea M, Bar-Dayan Y, Froy O. Influences of Breakfast on Clock Gene Expression and Postprandial Glycemia in Healthy Individuals and Individuals With Diabetes: A Randomized Clinical Trial. Diabetes Care. 2017 Nov;40(11):1573-1579. doi: 10.2337/dc16-2753. Epub 2017 Aug 22. PMID 28830875